CLINICAL TRIAL: NCT06056336
Title: Perioperative Immunoagent (Tislelizumab) Plus Chemotherapy for Locally Advanced Resectable Thoracic Oesophageal Squamous Cell Carcinoma Trail:A Prospective Single-arm,Phase II Study (PILOT Trail)
Brief Title: Perioperative Tislelizumab Plus Chemotherapy for Resectable Thoracic Oesophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guo Xufeng (Other)
Responsible Party: Sponsor-Investigator, Guo Xufeng, Principal Investigator, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS23059
Record Dates: First submitted 2023-09-10; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Chemoimmunotherapy; Adjuvant Therapy
Keywords: esophageal Squamous Cell Carcinoma; neoadjuvant chemotherapy; neoadjuvant immunotherapy; adjuvant therapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adjuvant tislelizumab plus chemothearpy (Experimental): Tislelizumab：200mg d1, q3w × 2 cycles，up yo 1 year; Nad-paclitaxel 260 mg/m2 d1 q3w 2 cycles;carboplatin AUC = 5 d1, q3w × 2 cycles.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg q21d up to 1 year. Nad-paclitaxel 260 mg/m2, IV., every 3 weeks, 2-3 cycles. Carboplatin area under the curve = 5, IV., every 3 weeks, 2 cycles.
  Other Names: Albumin-bound Paclitaxel; Carboplatin

SUMMARY:
The purpose of this study is to analyze esophageal cancer patients who underwent neoadjuvant immunotherapy with chemotherapy followed by esophagectomy to determine whether additional adjuvant therapy is associated with improved survival outcomes.

DETAILED DESCRIPTION:
Eligiled patients with pathologically confirmed thoracic esophageal squamous cell carcinoma and at clinical T1b-3N1-3M0 or T3N0M0 according to the eighth edition of American Joint Committee on Cancer staging will be allocated to neoadjuvant immunotherapy (tislelizumab 200mg d1, q3w × 2 cycles ) and chemotherapy (nad-paclitaxel 260 mg/m2 d1 + carboplatin AUC = 5 d1, q3w × 2 cycles) treatment. Patients with resected (R0) were assigned to receive tislelizumab ( at a dose of 200 mg every 3 weeks for 30 weeks) in pCR patients or adjuvant immunotherapy and chemothearpy for two cycles, and then tislelizumab ( at a dose of 200 mg every 3 weeks for 24 weeks) in non-pCR patients.The primary endpoint for this study is 2-year disease-free survival (DFS) in non-pCR patients.The secondary endpoints include pCR rate, major pathological response (MPR) rate, 2-year DFS in pCR patients, R0 resection rate, adverse events, and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteers to participate in the study, signs a consent form, has good compliance, and obeys the follow-up, and is willing and able to follow the protocol during the study;
2. Histologically-confirmed squamous cell carcinoma; tumors of the esophagus are located in the thoracic cavity;
3. Have not received systemic and local treatment for esophageal cancer;
4. Pre-treatment staging as cT1b-3N1-3M0 or T3N0M0, American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) 8th edition;
5. Male or female, aged ≥18 and ≤75 years;
6. The Eastern Cooperative Oncology Group (ECOG) performance status (PS) score is 0 -1;
7. R0 resection is expected;
8. Adequate cardiac function. All patients should perform electrocardiogram (ECG), and those with a cardiac history or ECG abnormality should perform echocardiography with the left ventricular ejection fraction >50%;
9. Adequate respiratory function with forced expiratory volume in 1 second (FEV1) ≥ 1.2 L, FEV1% ≥ 50% and lung diffusing capacity for carbon monoxide (DLCO) ≥ 50% shown in pulmonary function tests;
10. Adequate bone marrow function (white blood cells > 4×109/L, neutrophil > 1.5 ×109/L, hemoglobin > 90g/L, platelets > 100×109/L). Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3× upper level of normal (ULN);
11. Adequate liver function (total bilirubin <1.5× ULN, AST and ALT <2.5× ULN);
12. Adequate renal function (glomerular filtration rate (GFR) >60 mL/min; serum creatinine (SCr) ≤120 μmol/L];
13. Fertile female subjects are required to have a negative serum or urine pregnancy test no later than 72 hours before starting the study drug administration, and to use effective contraception (such as an IUD, contraceptive pill, or condom) during the trial period and for at least 3 months after the last dose; For male subjects whose partners are women of reproductive age, effective contraception should be used during the trial period and within 3 months after the last dose.

Exclusion Criteria:

1. Unresectable factors, including those who are unresectable for tumor reasons or have surgical contraindications, or who refuse surgery;
2. Patients with supraclavicular lymph node metastasis;
3. Poor nutritional status, BMI<18.5Kg/m2; Patients could continue to be considered for enrollment if corrected with symptomatic nutritional support before enrollment and after assessment by the principal investigator
4. Allergy to any drugs;
5. Have received or are receiving any of the following treatments; a) any radiotherapy, chemotherapy or other antineoplastic drugs directed at the tumour; b) being treated with an immunosuppressive drug or systemic hormone for immunosuppression (at a dose of >10mg/ day of prednisone or equivalent) within 2 weeks before the first dose of the study drug; Inhaled or topical steroids and corticosteroid replacement at doses >10mg/ day of prednisone or equivalent were allowed in the absence of active autoimmune disease; c) received live attenuated vaccine within 4 weeks before the first dose of study drug; d) major surgery or severe trauma within 4 weeks before the first dose of study drug;
6. Human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) active infection or known HIV seropositivity; including HBV or HCV surface antigen positive (RNA)
7. Uncontrolled cardiac symptoms or diseases, including but not limited to: (1) heart failure above NYHA class II, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias without or poorly controlled after clinical intervention;
8. Severe infection (CTCAE>2) occurred within 4 weeks before the first dose of study drug, such as severe pneumonia requiring hospitalization, bacteremia, and infectious complications; Prophylactic antibiotics were excluded if there was active pulmonary inflammation on chest imaging at baseline, if there were signs and symptoms of infection within 14 days before the first dose of the study drug, or if treatment with oral or intravenous antibiotics was required
9. Participation in other drug clinical studies within 4 weeks before randomization;
10. Patients with interstitial pneumonia or interstitial lung disease, or previous history of interstitial pneumonia or interstitial lung disease requiring hormone therapy, or other subjects with pulmonary fibrosis, organized pneumonia (such as bronchiolitis obliterans), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia that may interfere with the judgment and treatment of immune related pulmonary toxicity, or subjects with active pneumonia or severe lung function damage revealed by CT during screening; Active pulmonary tuberculosis;
11. Patients with any active autoimmune disease or history of autoimmune disease and possible recurrence [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients who can be controlled only by hormone replacement therapy can be enrolled)]; Patients with skin diseases that do not require systemic treatment, such as leukoplakia, psoriasis, alopecia, patients with type I diabetes that can be controlled by insulin treatment, or patients with a history of asthma, but have completely relieved in childhood and do not need any intervention, can be enrolled; Asthma patients who needed bronchodilators for intervention could not be enrolled; Patients have previously received an anti-PD-1，PD-L1 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways;
12. Other malignancies that had been diagnosed within 5 years before the first dose of a study drug were considered unless cancers with a low risk of metastasis or death (5-year survival rate, >90%), such as adequately treated basal-cell or squamous-cell skin cancer or carcinoma in situ of the cervix, were considered.
13. Pregnant or lactating women;
14. The investigators determined that there were other factors that might have led to the forced discontinuation of the study, such as other serious medical conditions (including mental illness) requiring co-treatment, alcohol, substance abuse, family or social factors, and factors that might have affected the safety or adherence of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival in non-pCR patients | Disease free survival time for recurrence or death within 2 years of surgery
  The time from the first day of surgery to the first occurrence of local or distant recurrence and metastasis or death from any cause in non-pCR patients

SECONDARY OUTCOMES:
pCR rate | 4 weeks after surgery
  Pathological complete response (pCR) rate of all patients
major pathological response | 4 weeks after surgery
  MPR was defined as the presence of viable tumor cells≤10% in the resected tumor specimen
2-year DFS in pCR patients | Disease free survival time for recurrence or death within 2 years of surgery
  The time from the first day of surgery to the first occurrence of local or distant recurrence and metastasis or death from any cause in pCR patients
R0 resection rate | 4 weeks after surgery
  No vital tumor is presented at the proximal, distal, or circumferential resection margin, then it is considered R0 resection
adverse events | Up to 100 months
  Safety will be evaluated for all treated patients using CTCAE V 5.0.
overall survival | Up to 5 years
  The date of death of any causes since the date of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Pan, Study Chair — the International Committee of Medical Journal Editors
Locations (1):
- Shanghai chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008
- [Result] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J. Long-term Efficacy of Neoadjuvant Chemoradiotherapy Plus Surgery for the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: The NEOCRTEC5010 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):721-729. doi: 10.1001/jamasurg.2021.2373. PMID 34160577
- [Result] Oppedijk V, van der Gaast A, van Lanschot JJ, van Hagen P, van Os R, van Rij CM, van der Sangen MJ, Beukema JC, Rutten H, Spruit PH, Reinders JG, Richel DJ, van Berge Henegouwen MI, Hulshof MC. Patterns of recurrence after surgery alone versus preoperative chemoradiotherapy and surgery in the CROSS trials. J Clin Oncol. 2014 Feb 10;32(5):385-91. doi: 10.1200/JCO.2013.51.2186. Epub 2014 Jan 13. PMID 24419108

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT06056336/Prot_SAP_000.pdf